CLINICAL TRIAL: NCT02609386
Title: A Randomized Phase 2 Trial of Neoadjuvant and Adjuvant Therapy With the IRX 2 Regimen in Patients With Newly Diagnosed Stage II, III, or IVA Squamous Cell Carcinoma of the Oral Cavity
Brief Title: IRX-2 Regimen in Patients With Newly Diagnosed Stage II, III, or IVA Squamous Cell Carcinoma of the Oral Cavity
Acronym: INSPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brooklyn ImmunoTherapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRX-2 2015-A
Record Dates: First submitted 2015-09-10; First posted 2015-11-20 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
Keywords: Head and Neck Neoplasms; Immunotherapy; Cancer; Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Neoplasms | interventions — IRX 2; Immunotherapy; Cyclophosphamide; Indomethacin; Anti-Inflammatory Agents, Non-Steroidal; Zinc; Geritol; Omeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen 1 (Experimental): IRX Regimen with IRX-2, cyclophosphamide, indomethacin, zinc-containing multivitamin, and omeprazole as neoadjuvant and adjuvant therapy.
  Interventions: Biological: IRX-2; Drug: Cyclophosphamide; Drug: Indomethacin; Dietary Supplement: Zinc-containing multivitamin; Drug: Omeprazole
- Regimen 2 (Active Comparator): Regimen 1 but without IRX-2
  Interventions: Drug: Cyclophosphamide; Drug: Indomethacin; Dietary Supplement: Zinc-containing multivitamin; Drug: Omeprazole

INTERVENTIONS:
Biological: IRX-2 — Method of Administration: Administered for 10 days as subcutaneous bilateral injections in the upper neck.
  Other Names: Immunotherapy
  Arms: Regimen 1
Drug: Cyclophosphamide — Method of Administration: Cyclophosphamide is administered once by IV
  Other Names: Cytophosphane; Cytoxan
Drug: Indomethacin — Method of Administration: Indomethacin is administered orally for 21 days.
  Other Names: NSAID; Indocin
Dietary Supplement: Zinc-containing multivitamin — Method of Administration: Zinc-containing multivitamin is administered orally for 21 days.
  Other Names: Zinc; Multi-vitamin
Drug: Omeprazole — Method of Administration: Omeprazole is administered orally for 21 days
  Other Names: Proton pump inhibitor; Prilosec

SUMMARY:
The purpose of this study is to determine whether a pre-operative regimen of the study drug, IRX-2, a human cell-derived biologic with multiple active cytokine components, plus a single dose of cyclophosphamide, followed by 21 days of indomethacin, zinc-containing multivitamins, and omeprazole is active in treatment of oral cavity cancer. The regimen is intended to stimulate an immune response against the cancer.

DETAILED DESCRIPTION:
This study will assess the activity and safety of the IRX Regimen in participants with newly diagnosed, untreated, surgically resectable squamous cell cancer of the oral cavity. Participants will be randomly assigned to receive either Regimen 1: IRX-2 + cyclophosphamide + indomethacin + zinc + omeprazole, or Regimen 2: cyclophosphamide + indomethacin + zinc + omeprazole.

The primary study hypothesis is that the Regimen 1 with IRX-2 prolongs event-free survival and overall survival when compared to Regimen 2 without IRX-2.

Subjects will be randomized to either Regimen 1 or Regimen 2 on a 2:1 basis and treated prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed (histology or cytology) clinical Stage II, III, or IVA squamous cell cancer of the oral cavity (excluding lip). Subjects must be staged using AJCC Cancer Staging Manual Edition 7.0 (appendices 1 and 2).
2. Disease surgically resectable with curative intent
3. Hematological function: hemoglobin >9 g/dL; lymphocyte count >0.50 x 109/L; neutrophil count >1.5 x 109/L; platelet count >100 x 109/L
4. Hepatic function: serum albumin >3.0 g/dL; aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <3x the upper limits of normal (ULN); alkaline phosphatase <2x the ULN
5. Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.4x the ULN
6. Calculated creatinine clearance > 50 mL/minute (Appendix 4)
7. At least 18 years of age
8. Willing and able to give informed consent and adhere to protocol therapy
9. Karnofsky performance status (KPS) >=70%
10. Females of childbearing potential (not surgically sterile or less than 12 months post-menopausal) must be able and willing to use a highly effective form of pregnancy prevention from the time of screening, during the study and 30 days after last dose of study regimen. Males with a partner of childbearing potential must use condoms with spermicide from the date of screening to 30 days after their last dose of study regimen
11. Negative urine/serum pregnancy test, if applicable

Exclusion Criteria:

1. Prior surgery, radiation therapy, or chemotherapy other than biopsy or emergency procedure required for supportive care of this oral cavity cancer.
2. Any medical contraindications or previous therapy that would preclude treatment with either IRX 2 Regimen 1 or 2 or the surgery, reconstruction or adjuvant therapy required to treat the oral tumor appropriately

   * Live vaccines should ideally not be administered to any patients undergoing treatment with chemotherapy or immunotherapy, but if need be, they should be administered >4 months prior to the initiation of treatment or >4 months after the completion of all treatment
   * Inactivated vaccines should precede the initiation of any study regimen and/or standard adjuvant therapy by at least 2 weeks, but preferably 4 weeks or longer
3. Clinical status of either subject or tumor such that administration of 21 day neoadjuvant IRX-2 Regimen 1 or 2 before surgery would be medically inappropriate
4. Tumor of the oropharynx
5. Tumor involvement of the following sites or any of these signs or symptoms likely to be associated with T4b cancer:

   * involvement of pterygopalatine fossa, maxillary sinus, or facial skin;.
   * gross extension of tumor to the skull base;
   * pterygoid plate erosion;
   * sphenoid bone or foramen ovale involvement;
   * direct extension to involve prevertebral fascia;
   * extension to superior nasopharynx or Eustachian tube;
   * direct extension into the neck with involvement of the deep neck musculature (neck node fixation);
   * suspected invasion (encasement) of the common or internal carotid arteries. Encasement will be assessed radiographically and will be defined as tumor surrounding the carotid artery 270º or greater;
   * direct extension of neck disease to involve the external skin;
   * direct extension to mediastinal structures;
   * regional metastases to the supraclavicular neck (low level IVB or VB)
6. Any investigational agent within the previous 30 days.
7. Daily administration of systemic immunosuppressive therapy or corticosteroids (except in physiological doses for hormone deficiency) during the previous 30 days.
8. Chronic anticoagulation, not including aspirin, but including heparins, warfarin, oral anticoagulation or other platelet function inhibitors, that can not, in the documented opinion of the investigator, safely be interrupted from at least 2 days prior to the initiation of the study regimen until after surgical resection of the tumor.
9. Symptomatic cardiopulmonary disease (including congestive heart failure and hypertension), coronary artery disease, serious arrhythmia or chronic lung disease. Patients with these conditions who are stable with relatively minor symptoms and who are appropriate candidates for surgical treatment of their tumor need not be excluded
10. Myocardial infarction within the last 3 months
11. Distant metastases (M1 disease).
12. Known infection with hepatitis B, hepatitis C, or HIV.
13. Signs or symptoms of systemic bacterial infection (use of antibiotics to treat superficial infection or contamination of tumor shall not, by itself, be considered evidence of infection).
14. Clinically significant gastritis or peptic ulcer disease that would contraindicate the use of indomethacin.
15. Stroke or other symptoms of cerebral vascular insufficiency within the last 3 months.
16. Allergy to ciprofloxacin (or other quinolones), acetylsalicylic acid, or indomethacin.
17. Previous diagnosis of invasive cancer from which the individual is NOT disease-free AND that has required treatment within the past 5 years, except for superficial skin, cervical cancer in-situ, well-differentiated thyroid or early stage prostate or bladder cancer (i.e., treatment with curative intent and long term disease-free expectations).
18. Prior axillary dissection.
19. Breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory T Wolf, MD, FACS, Principal Investigator — University of Michigan Hospitals
Locations (22):
- United States (13):
  - Banner University Medical Center, Tucson, Arizona
  - University of Arkansas For Medical Sciences, Little Rock, Arkansas
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Emory University - Winship Cancer Center, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Monter Cancer Center - North Shore LIJ, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Providence Cancer Center, Portland, Oregon
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
- Brazil (7):
  - Hospital Erasto Gaertner, Curitiba
  - Instituto Goiano de Oncologia e Hematologia (INGOH), Goiânia
  - Instituto do Câncer de Londrina, Londrina
  - Instituto Nacional do Cancer (INCA), Rio de Janeiro
  - Hospital de Base de São José do Rio Preto, São José do Vale do Rio Preto
  - Instituto Brasileiro de Controle do Câncer, São Paulo
  - Instituto do Cancer do Estado de São Paulo - ICESP, São Paulo
- Sunnybrook Research Institute, Toronto, Canada
- Queen Elizabeth University Hospital Glasgow, Glasgow, United Kingdom

REFERENCES:
- [Background] Wolf GT, Fee WE Jr, Dolan RW, Moyer JS, Kaplan MJ, Spring PM, Suen J, Kenady DE, Newman JG, Carroll WR, Gillespie MB, Freeman SM, Baltzer L, Kirkley TD, Brandwein HJ, Hadden JW. Novel neoadjuvant immunotherapy regimen safety and survival in head and neck squamous cell cancer. Head Neck. 2011 Dec;33(12):1666-74. doi: 10.1002/hed.21660. Epub 2011 Jan 31. PMID 21284052
- [Background] Berinstein NL, Wolf GT, Naylor PH, Baltzer L, Egan JE, Brandwein HJ, Whiteside TL, Goldstein LC, El-Naggar A, Badoual C, Fridman WH, White JM, Hadden JW. Increased lymphocyte infiltration in patients with head and neck cancer treated with the IRX-2 immunotherapy regimen. Cancer Immunol Immunother. 2012 Jun;61(6):771-82. doi: 10.1007/s00262-011-1134-z. Epub 2011 Nov 6. PMID 22057678
- [Derived] Wolf GT, Liu S, Bellile E, Sartor M, Rozek L, Thomas D, Nguyen A, Zarins K, McHugh JB; INSPIRE Trial Clinical Investigators. Tumor infiltrating lymphocytes after neoadjuvant IRX-2 immunotherapy in oral squamous cell carcinoma: Interim findings from the INSPIRE trial. Oral Oncol. 2020 Dec;111:104928. doi: 10.1016/j.oraloncology.2020.104928. Epub 2020 Jul 29. PMID 32738599
- See also: Sponsor's website — http://irxtherapeutics.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen 1: IRX Regimen with IRX-2, cyclophosphamide, indomethacin, zinc-containing multivitamins, and omeprazole as neoadjuvant and adjuvant therapy.
  IRX-2: Method of Administration: Administered for 10 days as subcutaneous bilateral injections in the upper neck.
  Cyclophosphamide: Method of Administration: Cyclophosphamide is administered once by IV
  Indomethacin: Method of Administration: Indomethacin is administered orally for 21 days.
  Zinc-containing multivitamins: Method of Administration: Zinc-containing multivitamin is administered orally for 21 days.
  Omeprazole: Method of Administration: Omeprazole is administered orally for 21 days.
- Regimen 2: Regimen 1 but without IRX-2.
  Cyclophosphamide: Method of Administration: Cyclophosphamide is administered once by IV
  Indomethacin: Method of Administration: Indomethacin is administered orally for 21 days.
  Zinc-containing multivitamin: Method of Administration: Zinc-containing multivitamins are administered orally for 21 days.
  Omeprazole: Method of Administration: Omeprazole is administered orally for 21 days.
Period: Overall Study
Arm/Group | Regimen 1 | Regimen 2
Started | 70 | 35
Completed | 42 | 18
Not Completed | 28 | 17
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Death | 19 | 9
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Regimen 1: IRX Regimen with IRX-2, cyclophosphamide, indomethacin, zinc-containing multivitamins, and omeprazole as neoadjuvant and adjuvant therapy.
  IRX-2: Method of Administration: Administered for 10 days as subcutaneous bilateral injections in the upper neck.
  Cyclophosphamide: Method of Administration: Cyclophosphamide is administered once by IV.
  Indomethacin: Method of Administration: Indomethacin is administered orally for 21 days.
  Zinc-containing multivitamins: Method of Administration: Zinc-containing multivitamins are administered orally for 21 days.
  Omeprazole: Method of Administration: Omeprazole is administered orally for 21 days
- Regimen 2: Regimen 1 but without IRX-2.
  Cyclophosphamide: Method of Administration: Cyclophosphamide is administered once by IV.
  Indomethacin: Method of Administration: Indomethacin is administered orally for 21 days.
  Zinc-containing multivitamins: Method of Administration: Zinc-containing multivitamins are administered orally for 21 days.
  Omeprazole: Method of Administration: Omeprazole is administered orally for 21 days.
- Total: Total of all reporting groups
Arm/Group | Regimen 1 | Regimen 2 | Total
Number analyzed (Participants) | 70 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.80) | 59.9 (11.50) | 59.7 (10.34)
Age, Continuous [Median (Full Range); unit: years] | 60.5 [38 to 81] | 61 [23 to 79] | 61 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 10 | 32
  Male | 48 | 25 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 12 | 40
  Not Hispanic or Latino | 41 | 22 | 63
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 58 | 25 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 0 | 2
  United States | 43 | 24 | 67
  Brazil | 24 | 11 | 35
  United Kingdom | 1 | 0 | 1
Primary Disease Stage [Count of Participants; unit: Participants] — Participants had their cancer staged using the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Edition 7. Staging is based on size of primary tumor, whether there is involvement in the lymph nodes, and the presence of distant metastatic disease.
  Participants with Stage I/II disease did not have any involvement in the lymph nodes or distant metatstatic disease. Participants with stage III/IV disease (more advanced disease) had a primary tumor >4 cm in greatest dimension with nodal involvement in at least one lymph node or mestatatic disease.
  Participants
    Primary disease Stage I/II | 26 | 11 | 37
    Primary disease Stage III/IV | 44 | 24 | 68

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)- Number of Participants With an Event
Description: EFS is defined as the time from randomization until progression after surgery, or at surgery, if failure to resect gross disease, or at time of death from any cause after randomization.
Time Frame: From randomization up until the data cut-off date of June 2, 2022 (approximately 76 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 | Regimen 2
Number analyzed (Participants) | 70 | 35
Participants | 31 | 15

2. Primary Outcome: EFS- Time to Event
Description: EFS is defined as the time from randomization until progression after surgery, or at surgery, if failure to resect gross disease, or at time of death from any cause after randomization. Assessment of progression/disease recurrence occurred by physical exam and annual imaging for the duration of the follow up portion of the study. Median EFS was estimated using the Kaplan-Meier method.
Time Frame: From randomization up until the data cut-off date of June 2, 2022 (approximately 76 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Regimen 1 | Regimen 2
Number analyzed (Participants) | 70 | 35
Months | 48.3 [11.4 to NA] — The upper limit for median EFS was not estimated because it was longer than the latest censoring time, and therefore was not achieved | NA [18.8 to NA] — Median EFS is not reported for the Regimen 2 population because it was not reached.The upper limit for median EFS was not estimated because it was longer than the latest censoring time, and therefore was not achieved.
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2; Test type: Other; p = 0.6176, Log Rank; Cox Proportional Hazard = 1.102, 95% CI 2-sided [0.6 to 2.1]

3. Secondary Outcome: Overall Survival (OS)- Number of Participants With an Event
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: From randomization up until the data cut-off date of June 2, 2022 (approximately 76 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 | Regimen 2
Number analyzed (Participants) | 70 | 35
Participants | 19 | 11
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2; Test type: Other; p = 0.3889, Log Rank; Cox Proportional Hazard = 1.009, 95% CI 2-sided [0.5 to 2.2]

4. Secondary Outcome: OS- Time to Event
Description: OS was defined as the time from randomization to death due to any cause. Data for partipants who were alive at the end of the study were censored at the last known alive date. Median OS was estimated using the Kaplan-Meier method.
Time Frame: From randomization up until the data cut-off date of June 2, 2022 (approximately 76 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Regimen 1 | Regimen 2
Number analyzed (Participants) | 70 | 35
Months | NA [NA to NA] — Median OS was not estimated because it was longer than the latest censoring time, and therefore was not achieved. In other words, there was an insufficient number of participants with events to calculate median OS, and the lower and upper limits of the 95% confidence interval | NA [42.6 to NA] — Median OS (and upper 95% CI) was not estimated because it was longer than the latest censoring time, and therefore was not achieved. In other words, there was an insufficient number of participants with events to calculate median OS and the upper limit of the 95% confidence interval
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2; Test type: Other; p = 0.5091, Log Rank; Cox Proportional Hazard = 1.009, 95% CI 2-sided [0.5 to 2.2]

ADVERSE EVENTS:
Time Frame: AEs/SAEs were collected over a period of approximately 60 days (i.e., from the day of randomization through 30 days after the last dose of study drug). If booster treatments were administered, AEs/SAEs were collected through 30 days after the last dose of study drug. AE data were collected over a period of approximately 2 years and 10 months. All cause mortality was assessed through study completion, approximately 76 months.
Description: # of participants at risk for all-cause mortality (70) differs from # at risk for serious and other AEs in Regimen 1 (68) as the population assessed for all-cause mortality was the intent to treat (ITT) population, i.e., all randomized subjects whether or not they received any component of the regimen they were randomized to. # of participants at risk for AE/SAEs (68) corresponds to the safety population, i.e., all pts who received at least 1 dose of study regimen.
Groups:
- Regimen 2: Regimen 1 but without IRX-2
  Cyclophosphamide: Method of Administration: Cyclophosphamide is administered once by IV.
  Indomethacin: Method of Administration: Indomethacin is administered orally for 21 days.
  Zinc-containing multivitamins: Method of Administration: Zinc-containing multivitamins are administered orally for 21 days.
  Omeprazole: Method of Administration: Omeprazole is administered orally for 21 days.
Arm/Group | Regimen 1 | Regimen 2
All-Cause Mortality (participants affected / at risk) | 19/70 | 11/35
Serious Adverse Events (participants affected / at risk) | 29/68 | 14/35
Other Adverse Events (participants affected / at risk) | 65/68 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (N=68) | Regimen 2 (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Salivary gland fistula (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oral cavity fistula (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Disease Progression (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Postoperative wound infection (Infections and infestations) | 4 | 2
Abscess neck (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 3 | 0
Lung infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 0
Graft ischaemia (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell count increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 2 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 2 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Venous haemorrhage (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (N=68) | Regimen 2 (N=35)
Anaemia (Blood and lymphatic system disorders) | 11 | 5
Atrial fibrillation (Cardiac disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 17 | 9
Nausea (Gastrointestinal disorders) | 15 | 6
Dry mouth (Gastrointestinal disorders) | 10 | 6
Constipation (Gastrointestinal disorders) | 10 | 4
Diarrhoea (Gastrointestinal disorders) | 12 | 2
Dysphagia (Gastrointestinal disorders) | 8 | 3
Oral pain (Gastrointestinal disorders) | 8 | 3
Vomiting (Gastrointestinal disorders) | 7 | 2
Glossodynia (Gastrointestinal disorders) | 5 | 0
Odynophagia (Gastrointestinal disorders) | 3 | 2
Oral cavity fistula (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 10 | 4
Injection site pain (General disorders) | 5 | 0
Face oedema (General disorders) | 4 | 0
Pyrexia (General disorders) | 0 | 3
Radiation skin injury (Injury, poisoning and procedural complications) | 12 | 4
Procedural pain (Injury, poisoning and procedural complications) | 4 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 4 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 2
Weight decreased (Investigations) | 14 | 6
Neutrophil count decreased (Investigations) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Headache (Nervous system disorders) | 6 | 4
Dysgeusia (Nervous system disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1
Lymphoedema (Vascular disorders) | 4 | 3

LIMITATIONS AND CAVEATS:
One of the initial secondary objectives of the study was to compare the feasibility of each booster regimen (Regimen 1 vs Regimen 2) post-surgery. However, as a significant number of patients were unable to receive booster treatments due to tolerability issues and/or their post-surgery/post-adjuvant chemoradiation therapy status, booster regimens were discontinued and analysis of booster feasibility was not performed due to insufficient data for a meaningful, statistically sound analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have the right to first publication. Following first publication, the Institution and/or Principal Investigator may publish data or results from the Study; provided, however, that the Institution and/or Principal Investigator submits the proposed publication to Sponsor for review at least 60 days prior to the date of the proposed publication. Sixty days shall be extended to 120 days if Sponsor determines that the publication contains patentable matter.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT02609386/Prot_SAP_000.pdf